CLINICAL TRIAL: NCT03816423
Title: The Use of Videos for Informed Consent for Prenatal Genetic Screening: a Randomized Controlled Trial
Brief Title: Use of Videos to Improve Patient Knowledge on Prenatal Genetics
Acronym: VPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00035994
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-03

CONDITIONS: Aneuploidy; Birth Defect
Keywords: patient education; genetic counseling
MeSH Terms: conditions — Aneuploidy; Congenital Abnormalities | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Primary purpose: assess and compare patient knowledge on prenatal genetic screening before and after a standard prenatal care visit compared to the addition of a pre-appointment educational video.
  All participants will complete a 15-item questionnaire on prenatal genetic screening options at baseline and after routine prenatal care visit.
  Participants randomized to the control group, will have a routine prenatal care appoinment, while the intervention group will watch a pre-appointment 4.5 minute educational video entitled "How to decide about prenatal genetic testing".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional counseling (No Intervention): Patients will undergo routine prenatal care visit with clinical practicioner only
- video group (Experimental): Participants randomized to the intervention group (video education) will view the prenatal screening video "How to Decide About Prenatal Genetic Testing," followed by a routine prenatal appointment.
  Interventions: Other: video

INTERVENTIONS:
Other: video — Participants randomized to the intervention group, will wacth a pre-appointment video, followed by a routine prenatal care visit.
  Arms: video group

SUMMARY:
This is a randomized controlled trial of a low income and low health literacy population of pregnant women from a diverse racial and ethnic background to assess the effectiveness of a pre-visit educational video on prenatal genetic screening and testing options.

DETAILED DESCRIPTION:
During pregnancy, women are routinely counseled about the risks of their offspring to have a chromosomal abnormality or birth defects. Both prenatal screening and diagnostic testing options to exclude aneuploidy should be offered to all pregnant women early in their pregnancy. A standardized educational video on prenatal screening may enhance a patient's understanding and knowledge of testing and support more informed decisions.

The objective of this study is to evaluate and compare patient knowledge scores on prenatal genetic screening before and after a standard prenatal care visit compared to the addition of a pre-appointment educational video.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy, english or spanish-speaking

Exclusion Criteria:

* minors <18 years old,
* > 21 completed weeks of gestational age,
* prior genetic counseling during current pregnancy
* fetus with known ultrasound abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Knowledge score | same day for both groups
  Evaluate the participants' baseline and post-visit knowledge scores on prenatal genetic screening for both groups using the "Maternal Serum Screening Knowledge Score Questionnaire" (MSSKQ)
Knowledge score change | same day for both groups
  Compare the knowledge score change for both groups using the Maternal Serum Screening Knowledge Score Questionnaire" (MSSKQ)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Leavitt, MD, MPH, Principal Investigator — University of South Florida
Locations (1):
- Genesis Healthpark- TGH, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No